CLINICAL TRIAL: NCT03634657
Title: Wirksamkeit Additiver Strahlenschutzvorrichtungen Zwecks Reduzierung Der Ionisierenden Streustrahlung im Herzkatheterlabor
Brief Title: EffectivenesS of Additional X-ray PRotection dEviceS in Reducing Scattered Radiation in Radial interventiOn
Acronym: ESPRESSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tommaso Gori (Other)
Responsible Party: Sponsor-Investigator, Tommaso Gori, Director, Cardiac Catheterization Laboratory ; Director, Study center of Center for Cardiology, university hospital Mainz, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ESPRESSO
Record Dates: First submitted 2018-08-08; First posted 2018-08-16 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Exposure of Member of Staff to Medical Diagnostic X-Ray
Keywords: Scattered radiation; X-ray protection; Radiation in cath lab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plain X-ray protection shield (Active Comparator)
  Interventions: Radiation: Plain X-ray protection shield
- Protection shield & X-ray protective strips (Experimental)
  Interventions: Radiation: Protection shield & X-ray protective strips
- Protection shield & protective strips & patient cut-outs (Experimental)
  Interventions: Radiation: Protection shield & protective strips & patient cut-outs

INTERVENTIONS:
Radiation: Plain X-ray protection shield — Coronary angiography with mere X-ray protection shield
  Arms: Plain X-ray protection shield
Radiation: Protection shield & X-ray protective strips — Coronary angiography with X-ray protection shield & X-ray protective strips
  Arms: Protection shield & X-ray protective strips
Radiation: Protection shield & protective strips & patient cut-outs — Coronary angiography with X-ray protection shield & X-ray protective strips & X-ray protection patient cut-outs
  Arms: Protection shield & protective strips & patient cut-outs

SUMMARY:
This study evaluates the radiation exposure of scattered radiation for the interventionalist during coronary angiography using different X-ray protection materials, namely, an X-ray Screen without additional X-ray protection, an X-ray Screen with additional protective strips and an X-ray Screen with additional protective strips AND protective patient cut-outs.

ELIGIBILITY:
Inclusion Criteria:

* indication for coronary angiography

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Operator dose | Duration of coronary angiography of individuel patient, varies between approximately 5 minutes of radiation (easy access, exclusion coronary heart disease) and app. 3 hours (difficult and complex percutaneous coronary intervention).
  Dose of radiation measured

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Anadol R, Brandt M, Merz N, Knorr M, Ahoopai M, Geyer M, Krompiec D, Wenzel P, Munzel T, Gori T. Effectiveness of additional X-ray protection devices in reducing scattered radiation in radial intervention: the ESPRESSO randomised trial. EuroIntervention. 2020 Oct 23;16(8):663-671. doi: 10.4244/EIJ-D-19-00945. PMID 32338611
- [Derived] Anadol R, Brandt M, Merz N, Knorr M, Ahoopai M, Geyer M, Krompiec D, Wenzel P, Munzel T, Gori T. Effectiveness of additional X-ray protection devices in reducing Scattered radiation in radial interventions: protocol of the ESPRESSO randomised trial. BMJ Open. 2019 Jul 3;9(7):e029509. doi: 10.1136/bmjopen-2019-029509. PMID 31272982